CLINICAL TRIAL: NCT05467995
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of AK111 in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Evaluate the Efficacy and Safety of AK111 in Subjects With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-202
Record Dates: First submitted 2022-02-10; First posted 2022-07-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Ankylosing Spondylitis
Keywords: AK111; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AK111 75mg (Experimental): AK111 75mg will be administered by subcutaneous injection at Week 0, 1 and 4 , followed by dosing every 4 weeks until Week12.
  Interventions: Biological: AK111
- AK111 150mg (Experimental): AK111 150mg will be administered by subcutaneous injection at Week 0, 1 and 4 , followed by dosing every 4 weeks until Week12.
  Interventions: Biological: AK111
- AK111 300mg (Experimental): AK111 300mg will be administered by subcutaneous injection at Week 0, 1 and 4 , followed by dosing every 4 weeks until Week12.
  Interventions: Biological: AK111
- Placebo (Placebo Comparator): Placebo will be administered by subcutaneous injection at Week 0, 1 and 4 , followed by dosing every 4 weeks until Week12.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AK111 — AK111 administered subcutaneously at Week 0, 1, and 4, then every 4 weeks
  Arms: AK111 150mg; AK111 300mg; AK111 75mg
Biological: Placebo — Placebo administered subcutaneously at Week 0, 1, and 4, then every 4 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of AK111 in subjects with active ankylosing spondylitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of AK111 in the treatment of subjects with active ankylosing spondylitis. Subjects will be randomized to receive AK111 or placebo following subcutaneous injection. The study period for each subject will be 25 weeks, including a screening period of up to 35 days, followed by a treatment period of 12 weeks and a follow up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years old.
* Ankylosing spondylitis has been diagnosed for at least 6 months before screening, with radiological evidence that meets the Modified New York Criteria for Ankylosing Spondylitis.
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 and Spinal pain score≥ 4 (based on BASDAI question 2).
* Subjects received at least 1 kind of non-steroidal anti-inflammatory drugs (NSAIDs), prior to randomization with an inadequate response or failure to respond.
* Subjects who are regularly taking NSAIDs, weak opioids or oral glucocorticoids as part of their AS therapy are required to be on a stable dose for at least 14 days before randomization.
* Subjects taking methotrexate (MTX) (≤25mg/week) or Sulfasalazine (≤3g/day) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 4 weeks before randomization.

Exclusion Criteria:

* Subjects with total ankylosis of the spine.
* Subjects with progressive or uncontrolled diseases of respiratory, circulatory, digestive, urogenital, endocrine, nervous or mental systems, or with other chronic diseases that are not suitable to participate to the study.
* Subjects with other inflammatory diseases or autoimmune diseases except Ankylosing spondylitis (AS).
* Subjects with any severe systemic or local infection within 2 months before screening.
* Subjects who are using strong opioid analgesics.
* Combined use of Disease Modifying Anti-Rheumatic Drugs (DMARDs) other than methotrexate and sulfasalazine, including but not limited to thalidomide, iguratimod, etc. within 4 weeks before randomization.
* Received any live vaccine within 2 months before screening or planned to receive any live vaccine during the study period.
* Previous exposure to secukinumab, ixekizumab or any other biologic drug directly targeting IL-17 or IL-17 receptor.
* Received Natalizumab or other drugs that regulate B cells or T cells within 6 months before screening.
* Received more than 2 kinds of Tumor necrosis factor alpha(TNF-α) inhibitors before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who achieve Assessment of SpondyloArthritis International Society 20% improvement (ASAS20) response at Week 16. | Week16
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global, pain, function (assessed by BASFI) and inflammation (mean of Ankylosing Spondylitis Disease Activity Index [BASDAI] question 5 and 6 ). ASAS20 response is defined as improvement of ≥ 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and ≥1 unit in the remaining domain.
Percentage of subjects with treatment-emergent adverse events (TEAEs) during the study. | Baseline to Week20
Percentage of subjects with treatment-emergent serious adverse events (SAEs) during the study. | Baseline to Week20

SECONDARY OUTCOMES:
Percentage of subjects who achieve SpondyloArthritis International Society 40% improvement (ASAS40) response at Week 16. | Week 16
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global, pain, function (assessed by BASFI) and inflammation (mean of Ankylosing Spondylitis Disease Activity Index [BASDAI] question 5 and 6 ). ASAS40 response is defined as improvement of ≥40% and ≥2 units in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening in the remaining domain.
Percentage of subjects who achieve ASAS20 response at each visit from baseline. | Baseline to Week 20
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global, pain, function (assessed by BASFI) and inflammation (mean of Ankylosing Spondylitis Disease Activity Index [BASDAI] question 5 and 6 ). ASAS20 response is defined as improvement of ≥ 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and ≥1 unit in the remaining domain.
Percentage of subjects who achieve ASAS40 at each visit from baseline. | Baseline to Week 20
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global, pain, function (assessed by BASFI) and inflammation (mean of Ankylosing Spondylitis Disease Activity Index [BASDAI] question 5 and 6 ). ASAS40 response is defined as improvement of ≥40% and ≥2 units in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening in the remaining domain.
Change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at each visit from baseline. | Baseline to Week 20
  The Ankylosing Spondylitis Quality of Life (ASQoL), a validated disease-specific 18-item questionnaire, has been developed specifically for measuring health-related quality of life (HRQoL) in subjects with ankylosing spondylitis (AS) . The ASQoL score ranges from 0 to 18 with a higher score indicating worse HRQoL.
pharmacodynamics(PD) parameters: Changes of Interleukin-17A (IL-17A) level in peripheral serum compared with baseline and its relationship with AK111 exposure. | Baseline to Week 20
Immunogenicity: Number and percentage of subjects with detectable anti-AK111 antibody (ADA). | Baseline to Week 20
Change from baseline on the 36-item Short-Form (SF-36) Health Survey at each visit from baseline. | Baseline to Week 20
  The SF-36 is a 36-item generic health status measure. It measures 8 general health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Each of the 8 domain scores and the component summary scores range from 0 to 100, with higher scores indicating better health status.
Area under the curve from 0 to the time of the last quantifiable concentration (AUC0-t) | Baseline to Week 20
Maximum observed concentration (Cmax) | Baseline to Week 20
Terminal elimination half-life (T1/2) | Baseline to Week 20
Time of occurrence of Cmax (Tmax) | Baseline to Week 20

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The first affiliated hospital of Bengbu medical college, Bengbu, Anhui
  - Peking university people's hospital, Beijing, Beijing Municipality
  - Peking University Shougang hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu hospital capital medical university, Beijing, Beijing Municipality
  - Guangdong provincial people's hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first Bethune hospital of Jilin university, Changchun, Jilin
  - Second hospital of Shanxi Medical university, Taiyuan, Shanxi
  - The seventh affiliated hospital, Sun Yat-sen university, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No